CLINICAL TRIAL: NCT03087708
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study of an Oral, Selective Peripheral Opioid Receptor Antagonist in Advanced Non-Small Cell Lung Cancer
Brief Title: Naloxegol in Treating Patients With Stage IIIB-IV Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A221504; NCI-2016-01503 (Registry Identifier: Clinical Trial Reporting Program)
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Results first posted 2022-08-03 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group I (lower dose naloxegol, placebo) (Active Comparator): Patients receive lower dose naloxegol PO QD and placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.
  Interventions: Drug: Naloxegol; Other: Placebo; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Group II (placebo, higher dose naloxegol) (Active Comparator): Patients receive placebo PO QD and higher dose naloxegol PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.
  Interventions: Drug: Naloxegol; Other: Placebo; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Group III (placebo) (Placebo Comparator): Patients receive placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.
  Interventions: Other: Placebo; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Naloxegol — Given PO
  Arms: Group I (lower dose naloxegol, placebo); Group II (placebo, higher dose naloxegol)
Other: Placebo — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies the side effects and best dose of naloxegol and to see how well it works in treating patients with stage IIIB-IV non-small cell lung cancer. Naloxegol may relieve some of the side effects of opioid pain medication and fight off future growth in the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine feasibility and safety of long-term administration of two doses of a peripheral opioid receptor antagonist in patients with advanced non-small cell lung cancer (NSCLC) receiving first-line systemic therapy.

SECONDARY OBJECTIVES:

I. To explore whether patients randomized to one or both of the two study drug arms have less decline in health-related quality of life (HRQoL) than patients randomized to placebo.

II. To estimate the difference in the pain levels and opioid/non-opioid analgesic requirements between patients receiving naloxegol or placebo.

III. To estimate the difference in the adverse peripheral effects of opioids (e.g. constipation, nausea/emesis, dry mouth and urinary retention) between patients receiving naloxegol or placebo.

IV. To explore whether there is a signal that naloxegol may be associated with longer progression-free survival (PFS) and overall survival (OS).

V. To evaluate the difference in discontinuation rate of systemic therapy due to adverse events (AEs) and deaths attributable to systemic therapy.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (stage IIIB or IV) non-small cell lung cancer diagnosed by biopsy of the primary or metastatic site (American Joint Committee on Cancer 7.0)
* No known presence of known EGFR or EML4-ALK driver mutations in the tumor
* Started first-line systemic therapy of the investigator's choice within 12 weeks prior to registration, or planning to initiate first-line systemic therapy of the investigator's choice within 4 weeks after registration; no planned initiation of definitive (potentially curative) concurrent chemo-radiation
* No prior systemic therapy for advanced NSCLC, including chemotherapy, targeted therapy or immunotherapy (other than current treatment); prior palliative radiation permitted; prior adjuvant systemic therapy /radiation is permitted
* No more than 7 days of prior use of mixed opioid agonist/opioid antagonists or other opioid antagonists within 4 weeks before registration; patients should not receive such medications after registration and for the entire duration of study treatment
* No methadone within 4 weeks prior to registration
* Patients must have used opioid medication(s) for pain at some time in the 4 weeks prior to registration; current use of opioids (at the time of registration) and/or later during the course of the study is permitted but not required
* Expected survival > 3 months
* No concurrently active second invasive malignancies except non-melanoma skin cancer
* No history of gastrointestinal obstruction, or conditions that increase the risk of gastrointestinal obstruction, perforation, bleeding or impairment of the gastrointestinal wall; no abdominal surgery within 60 days of registration
* No acute gastrointestinal conditions, such as: obstruction, fecal impaction, obstipation, acute surgical abdomen, ongoing need for manual maneuvers to induce bowel movements (such as digital evacuation)
* No conditions that may compromise blood-brain barrier permeability (e.g., multiple sclerosis, recent brain trauma, Alzheimer's disease, or uncontrolled seizures)

  * No symptomatic and untreated brain metastases; patients will be eligible for study if radiation therapy for brain metastases was completed at least 7 days prior to registration
  * Patients having received stereotactic radiation will be eligible if the radiation was completed at least 7 days prior to registration
  * Patients having undergone surgical resection of brain metastases will be eligible after they have healed and recovered from the surgical intervention sufficiently to start systemic treatment for NSCLC, as determined by a neurosurgeon
  * No known leptomeningeal carcinomatosis
* No history of myocardial infarction =< 6 months prior to registration; no current symptomatic congestive heart failure, uncontrolled angina, or uncontrolled cardiac arrhythmias
* No severe hepatic impairment (Child-Pugh class C) or acute liver disease
* No known serious or severe hypersensitivity reaction to naloxegol or any of its excipients
* No concurrent use of moderate/strong CYP3A4 inhibitors, or strong CYP3A4 inducers
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown; therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required; a female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Calculated (calc.) creatinine clearance >= 60 mL/min calculated using the Cockcroft-Gault formula
* Total bilirubin =< 1.2 x upper limit of normal (ULN) unless due to Gilbert's disease
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Gupta, MD, Study Chair — Minneapolis VA Health Care System (University of Minnesota)
Locations (660):
- United States (660):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Middlesex Hospital, Middletown, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - South Florida Baptist Hospital, Plant City, Florida
  - Saint Anthony's Hospital Cancer Care Center, St. Petersburg, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Saint Claire Regional Medical Center, Morehead, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Beverly Hospital, Beverly, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kenansville, Kenansville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Scotland Memorial Hospital-Laurinburg Cancer Center, Laurinburg, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Vidant Oncology-Richlands, Richlands, North Carolina
  - WG Hefner VA Medical Center, Salisbury, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I (Lower Dose Naloxegol, Placebo): Patients receive lower dose naloxegol PO QD and placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.> > Naloxegol: Given PO>
  > Placebo: Given PO>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Quality-of-Life Assessment: Ancillary studies
- Group II (Placebo, Higher Dose Naloxegol): Patients receive placebo PO QD and higher dose naloxegol PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.> > Naloxegol: Given PO>
  > Placebo: Given PO>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Quality-of-Life Assessment: Ancillary studies
- Group III (Placebo): Patients receive placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.>
  > Placebo: Given PO>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Started | 17 | 16 | 17
Completed | 15 | 15 | 13
Not Completed | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Group I (Lower Dose Naloxegol, Placebo): Patients receive lower dose naloxegol PO QD and placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.>> >> Naloxegol: Given PO>>
  >> Placebo: Given PO>>
  >> Laboratory Biomarker Analysis: Correlative studies>>
  >> Quality-of-Life Assessment: Ancillary studies
- Group II (Placebo, Higher Dose Naloxegol): Patients receive placebo PO QD and higher dose naloxegol PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.>> >> Naloxegol: Given PO>>
  >> Placebo: Given PO>>
  >> Laboratory Biomarker Analysis: Correlative studies>>
  >> Quality-of-Life Assessment: Ancillary studies
- Group III (Placebo): Patients receive placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.>>
  >> Placebo: Given PO>>
  >> Laboratory Biomarker Analysis: Correlative studies>>
  >> Quality-of-Life Assessment: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo) | Total
Number analyzed (Participants) | 15 | 15 | 13 | 43
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.0 [57.0 to 71.0] | 67.0 [65.0 to 73.0] | 62.0 [60.0 to 67.0] | 66.0 [60.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 4 | 16
  Male | 6 | 12 | 9 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 12 | 41
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 12 | 11 | 12 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Planned use of Bevacizumab [Count of Participants; unit: Participants]
  No | 14 | 14 | 13 | 41
  Yes | 1 | 1 | 0 | 2
ECOG Performance Score [Count of Participants; unit: Participants] — Measure Description: ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction.
  ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0-1 | 10 | 12 | 11 | 33
    2 | 5 | 3 | 2 | 10
Pathologic T Stage [Count of Participants; unit: Participants] — Tx: Main tumor cannot be measured.
  T0: There is no evidence of a primary tumor.
  T1-T4 describe the size and location of the tumor. A larger tumor or a tumor that has grown deeper into nearby tissue will get a higher number and letter.
  From best to worst, T0, T1a, T1b, T2a, T2b, T3a, T3b, T4.
  Participants
    T0 | 0 | 1 | 0 | 1
    T1a | 0 | 2 | 0 | 2
    T1b | 2 | 1 | 2 | 5
    T2a | 2 | 2 | 1 | 5
    T2b | 1 | 1 | 1 | 3
    T3a | 2 | 2 | 2 | 6
    T3b | 0 | 2 | 0 | 2
    T4 | 5 | 0 | 5 | 10
    Tx | 3 | 4 | 2 | 9
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 6 | 4 | 8 | 18
  Former smoker (no smoking for one year or more) | 8 | 11 | 4 | 23
  Never smoked (less than 100 cigarettes in lifetime) | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Observed Accrual Rate Defined as Rate of Accrual Remaining >= 80% of the Expected
Description: Calculated as the total number of patients accrued to the study over two years divided by 184, the total expected accrual of patients evaluable for the primary endpoint.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Groups:
- Expected Accrued Patients: Expected accrued patients to be evaluable
Arm/Group | Expected Accrued Patients
Number analyzed (Participants) | 184
proportion of participants | 0.272

2. Primary Outcome: Proportion of Patients Alive Who Continue Study Drug and Complete the Health-related Quality of Life and Other Forms
Description: The proportion of patients alive at 6 months who continue study drug and complete the health-related quality of life and other forms for at least 6 months will be calculated by arm.
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: Ratio of patients evaluable for endpoint
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 15 | 15 | 13
Ratio of patients evaluable for endpoint | 0.4667 [0.2127 to 0.7341] | 0.4667 [0.2127 to 0.7341] | 0.3846 [0.1386 to 0.6842]

3. Primary Outcome: Incidence of Adverse Events as Described and Graded by the National Cancer Institute's Common Terminology Criteria for Adverse Events, Version 4.0
Description: The frequency of adverse events will be summarized by arm and compared between each treatment arm vs the placebo arm using Fisher's exact test. <3 is better and 3+ is worse.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Group I (Lower Dose Naloxegol, Placebo): Patients receive lower dose naloxegol PO QD and placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.> >>
  >
  >> Naloxegol: Given PO>
  >>
  >
  >> Placebo: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies
- Group II (Placebo, Higher Dose Naloxegol): Patients receive placebo PO QD and higher dose naloxegol PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.> >>
  >
  >> Naloxegol: Given PO>
  >>
  >
  >> Placebo: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies
- Group III (Placebo): Patients receive placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.>
  >>
  >
  >> Placebo: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 15 | 15 | 13
Participants
  Hematologic Adverse Events (regardless of attribution) : 3+ | 4 | 3 | 2
  Hematologic Adverse Events (regardless of attribution) : <3 | 11 | 12 | 11
  Non-Hematologic Adverse Events (regardless of attribution) : 3+ | 9 | 9 | 6
  Non-Hematologic Adverse Events (regardless of attribution) : <3 | 6 | 6 | 7
  Hematologic Adverse Events (at least possibly related to study) : 3+ | 1 | 0 | 0
  Hematologic Adverse Events (at least possibly related to study) : <3 | 14 | 15 | 13
  Non-Hematologic Adverse Events (at least possibly related to study) : 3+ | 1 | 3 | 0
  Non-Hematologic Adverse Events (at least possibly related to study) : <3 | 14 | 12 | 13
Statistical Analysis 1: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Comparison of Hematologic 3+ vs Hematologic <3; Test type: Other; p < 1, Fisher Exact
Statistical Analysis 2: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Comparison of Non-Hematologic 3+ vs Non-Hematologic <3; Test type: Other; p < 0.7051, Fisher Exact
Statistical Analysis 3: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Comparison of Hematologic 3+ vs Hematologic <3; Test type: Other; p < 0.6546, Fisher Exact
Statistical Analysis 4: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Comparison of Non-Hematologic 3+ vs Non-Hematologic <3; Test type: Other; p < 0.7051, Fisher Exact
Statistical Analysis 5: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Comparison of Non-Hematologic 3+ vs Non-Hematologic <3; Test type: Other; p < 0.2262, Fisher Exact
Statistical Analysis 6: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Comparison of Hematologic 3+ vs Hematologic <3; Test type: Other; p < 1, Fisher Exact
Statistical Analysis 7: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Comparison of Non-Hematologic 3+ vs Non-Hematologic <3; Test type: Other; p < 1, Fisher Exact

4. Secondary Outcome: Change in Trial Outcome Index
Description: Health-related quality of life scores at each timepoint and changes in scores between 6 months and baseline will be summarized by mean standard deviation, median (inter-quartile range). Scores will be plotted to explore the pattern over time and to examine differences between treatment arms. Differences in health-related quality of life between the treatment arms and the placebo arm will be conducted through linear mixed models and growth curve models to account for repeated assessments. Trial outcome index score is 0-92 with 0 being the worst and 92 being the best.
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Group I (Lower Dose Naloxegol, Placebo): Patients receive lower dose naloxegol PO QD and placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.
  >
  >
  >
  >
  >
  > Naloxegol: Given PO
  >
  >
  >
  >
  >
  > Placebo: Given PO
  >
  >
  >
  >
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  >
  >
  >
  >
  > Quality-of-Life Assessment: Ancillary studies
- Group II (Placebo, Higher Dose Naloxegol): Patients receive placebo PO QD and higher dose naloxegol PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.
  >
  >
  >
  >
  >
  > Naloxegol: Given PO
  >
  >
  >
  >
  >
  > Placebo: Given PO
  >
  >
  >
  >
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  >
  >
  >
  >
  > Quality-of-Life Assessment: Ancillary studies
- Group III (Placebo): Patients receive placebo PO QD. Courses repeat every 3 weeks in year 1 and then every 3 months in year 2 in the absence of unacceptable toxicity.
  >
  >
  >
  >
  >
  > Placebo: Given PO
  >
  >
  >
  >
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  >
  >
  >
  >
  > Quality-of-Life Assessment: Ancillary studies
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 7 | 7 | 5
units on a scale | 21.0 [0.0 to 27.0] | 14.0 [-4.0 to 20.0] | 9.0 [-1.0 to 10.0]

5. Secondary Outcome: Change in Function Subscales
Description: Health-related quality of life scores at each timepoint and changes in scores between 6 months and baseline will be summarized by mean standard deviation, median (inter-quartile range). Scores will be plotted to explore the pattern over time and to examine differences between treatment arms. Differences in health-related quality of life between the treatment arms and the placebo arm will be conducted through linear mixed models and growth curve models to account for repeated assessments. Function subscales score is 0-28 with 0 being the worst and 28 being the best.
Time Frame: Baseline to 6 months
Population: Two patients on the Naloxegol 12.5 mg arm did not complete all of the questions for the Fact-L at 6 months.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 7 | 7 | 5
units on a scale
  Physical Well Being: number analyzed (Participants) | 5 | 7 | 5
  Physical Well Being | 4.7 [3.0 to 8.0] | 0.0 [-3.0 to 3.0] | -0.3 [-5.8 to 0.0]
  Social Function Well Being: number analyzed (Participants) | 5 | 7 | 5
  Social Function Well Being | 6.0 [-3.0 to 9.0] | 5.0 [-2.0 to 7.0] | -2 [-3.0 to 1.0]
  Emotional Well Being: number analyzed (Participants) | 6 | 7 | 5
  Emotional Well Being | 2.5 [1.0 to 4.0] | 3.0 [0.0 to 7.0] | 0 [0.0 to 1.0]
  Functional Well Being: number analyzed (Participants) | 6 | 7 | 5
  Functional Well Being | 6.5 [2.0 to 8.0] | 5.0 [-3.0 to 10.0] | 4.0 [3.0 to 6.0]

6. Secondary Outcome: Change in Lung Cancer Subscale of the Functional Assessment of Cancer Therapy-Lung
Description: Health-related quality of life scores at each timepoint and changes in scores between 6 months and baseline will be summarized by mean standard deviation, median (inter-quartile range). Scores will be plotted to explore the pattern over time and to examine differences between treatment arms. Differences in health-related quality of life between the treatment arms and the placebo arm will be conducted through linear mixed models and growth curve models to account for repeated assessments. Lung cancer subscale score is 0-36 with 0 being the worst and 36 being the best.
Time Frame: Baseline to 6 months
Population: Two patients on the Naloxegol 12.5 mg arm did not complete all of the questions for the Fact-L at 6 months.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 6 | 7 | 5
units on a scale | 6.0 [-3.0 to 11.0] | 1.0 [0.0 to 6.0] | 1.0 [-2.0 to 6.0]

7. Secondary Outcome: Patient-reported Outcome Assessed by Patient-Reported Outcome-Common Terminology Criteria for Adverse Events
Description: Patient-Reported Outcome-Common Terminology Criteria for Adverse Events items will be summarized by arm. Patient-Reported Outcome-Common Terminology Criteria for Adverse Events response will be compared between the treatment arms vs. placebo arm using a chi-square test or Fisher's exact test as appropriate. Chosen PRO-CTCAE question is "In the last 7 days, what was the SEVERITY of your PAIN IN THE ABDOMEN (BELLY AREA) at its WORST?"
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 7 | 7 | 5
Participants
  None | 7 | 5 | 2
  Mild | 0 | 0 | 1
  Moderate | 0 | 2 | 1
  Missing | 0 | 0 | 1
Statistical Analysis 1: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Test type: Other; p < 0.68182, Fisher Exact
Statistical Analysis 2: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Test type: Other; p < 0.1091, Fisher Exact

8. Secondary Outcome: Patient-reported Outcome Assessed by a Urinary Retention Linear Analogue Self-Assessment
Description: Linear Analogue Self-Assessment items will be summarized by arm. Linear Analogue Self-Assessment scores will be compared between treatment arms versus placebo arm using Wilcoxon test. Linear Analogue Self-Assessment score is 0-10, with 0 being no trouble with ability to urinate easily and 10 being worst trouble with ability to urinate easily.
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 7 | 7 | 5
units on a scale | 0.0 [0.0 to 0.0] | 0.0 [-3.0 to 0.0] | 0.0 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Test type: Other; p < 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Test type: Other; p < 0.3339, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Opioid-induced Constipation Rating Scale
Description: Opioid-induced constipation rating scale will be summarized by arm. Scores will be compared between treatment arms vs. placebo arm using Wilcoxon test. Question from Bowel Function Diary is "In the past 24 hours, how much pain did you feel in your abdomen because of constipation?". Opioid-induced constipation rating scale is from 0-6, with 0 being none and 6 being very severe.
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 7 | 7 | 5
units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Test type: Other; p < 0.5930, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Test type: Other; p < 0.3105, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Level of Pain
Description: Pain scores will be summarized by arm. Pain scores will be compared between treatment arms vs. placebo using Wilcoxon test. Pain score scale is 0-10, with 10 being worst pain imaginable
Time Frame: Baseline to 6 months
Population: Only 19 patients completed the primary endpoint of staying on treatment and completing QOL booklets for 6 months.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 15 | 13 | 12
units on a scale
  Average Pain Scores at Baseline ( | 6.5 [5.0 to 8.0] | 5.0 [1.0 to 7.0] | 4.5 [4.0 to 7.0]
  Average Pain Scores at 6 Months: number analyzed (Participants) | 7 | 7 | 5
  Average Pain Scores at 6 Months | 0.0 [0.0 to 7.0] | 3.7 [0.0 to 6.0] | 2.2 [0.0 to 5.7]
Statistical Analysis 1: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Average Pain Scores at Baseline; Test type: Other; p = 0.6024, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Average Pain Scores at Baseline; Test type: Other; p < 0.3116, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Average Pain Scores at 6 Months; Test type: Other; p < 0.7712, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Average Pain Scores at 6 Months; Test type: Other; p < 1.0, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Analgesic Use
Description: The protocol-defined analysis for this secondary endpoint was not performed due to not specifying analgesic use in the questionnaire. Analgesic use will be summarized by arm. Frequencies of analgesic used will be compared using chi-square test or Fisher's exact test, as appropriate.
Time Frame: Up to 2 years
Population: Only 19 patients completed the primary endpoint of staying on treatment and completing QOL booklets for 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 15 | 13 | 12
Participants
  Analgesic use at Baseline?: Yes | 13 | 10 | 11
  Analgesic use at Baseline?: No | 2 | 3 | 1
  Analgesic use at Baseline?: Missing | 0 | 0 | 0
  Analgesic Use at 6 Months?: number analyzed (Participants) | 7 | 7 | 5
  Analgesic Use at 6 Months?: Yes | 3 | 5 | 2
  Analgesic Use at 6 Months?: No | 4 | 2 | 2
  Analgesic Use at 6 Months?: Missing | 0 | 0 | 1
Statistical Analysis 1: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Analgesic Use at 6 Months; Test type: Other; p < 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Analgesic Use at 6 Months; Test type: Other; p < 0.5758, Fisher Exact
Statistical Analysis 3: Comparison: Group I (Lower Dose Naloxegol, Placebo) vs Group III (Placebo); Analgesic use at Baseline; Test type: Other; p < 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Group II (Placebo, Higher Dose Naloxegol) vs Group III (Placebo); Analgesic use at Baseline; Test type: Other; p = 0.5930, Fisher Exact

12. Secondary Outcome: Unexpected Clinical Outcomes With Chemotherapy
Description: A Fisher's exact test was not performed due to low sample size. Frequency of discontinuation of chemotherapy will be summarized by arm and compared between each treatment arm vs the placebo arm using Fisher's exact test.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 17 | 16 | 17
Participants
  Treatment (Intervention) Completed Per Protocol Criteria | 2 | 1 | 2
  Patient Withdrawal/Refusal After Beginning Protocol Therapy (Intervention) | 3 | 5 | 6
  Adverse Events/Side Effects/Complications | 1 | 1 | 1
  Patient Off-Treatment (Intervention) For Other Complicating Disease | 1 | 0 | 0
  Death On Study | 2 | 6 | 4
  Other | 4 | 3 | 2
  Patient Withdrawal/Refusal Prior To Beginning Protocol Therapy (Intervention) | 2 | 0 | 2
  Missing | 2 | 0 | 0

13. Secondary Outcome: Progression-free Survival Assessed by Using the Standard Response Evaluation Criteria in Solid Tumors 1.1 Criteria
Description: Progression-free survival probabilities will be estimated by arm using the Kaplan-Meier estimator. In an exploratory manner, a Cox proportional hazards model will be used to determine the effect of naloxegol on progression-free survival.
Time Frame: From randomization to disease progression/relapse, death, or loss to follow-up, whichever occurs first, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 15 | 15 | 13
Participants
  Censored | 8 | 6 | 7
  Death | 5 | 4 | 1
  Progression | 2 | 5 | 5

14. Secondary Outcome: Overall Survival
Description: Overall survival probabilities will be estimated by arm using the Kaplan-Meier estimator. In an exploratory manner, a Cox proportional hazards model will be used to determine the effect of naloxegol on overall survival.
Time Frame: From randomization to death or loss to follow-up, whichever occurs first, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Naloxegol, Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group III (Placebo)
Number analyzed (Participants) | 15 | 15 | 13
Participants
  Censored | 9 | 6 | 7
  Death | 6 | 9 | 6

15. Other Pre Specified Outcome: Prognostic Effect of MOR Expression/Interaction on Health-related Quality of Life
Description: The protocol-defined analysis for this secondary endpoint was not performed due to being a correlative endpoint and not being collected in the data. MOR expression and activation will be included as a covariate in the linear mixed model, an interaction between MOR expression/activation and treatment will be evaluated.
Time Frame: Up to 2 years
Reporting Status: Not Posted, anticipated posting 2025-07

ADVERSE EVENTS:
Time Frame: 5 Years
Description: For Group I (Lower Dose Naloxegol, Placebo), 2 patients withdrew prior to starting treatment and no AE data was collected.
  For Group III (Placebo), 3 patients withdrew prior to starting treatment and no AE data was collected.
Arm/Group | Group III (Placebo) | Group II (Placebo, Higher Dose Naloxegol) | Group I (Lower Dose Naloxegol, Placebo)
All-Cause Mortality (participants affected / at risk) | 6/17 | 10/16 | 8/17
Serious Adverse Events (participants affected / at risk) | 7/14 | 9/16 | 9/15
Other Adverse Events (participants affected / at risk) | 13/14 | 11/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group III (Placebo) (N=14) | Group II (Placebo, Higher Dose Naloxegol) (N=16) | Group I (Lower Dose Naloxegol, Placebo) (N=15)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 3 (3) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Sudden death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group III (Placebo) (N=14) | Group II (Placebo, Higher Dose Naloxegol) (N=16) | Group I (Lower Dose Naloxegol, Placebo) (N=15)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 2 (14) | 3 (3)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (20) | 6 (16) | 4 (6)
Constipation (Gastrointestinal disorders) | 2 (10) | 0 (0) | 1 (13)
Diarrhea (Gastrointestinal disorders) | 5 (10) | 4 (9) | 4 (11)
Dry mouth (Gastrointestinal disorders) | 6 (26) | 3 (27) | 7 (12)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Flatulence (Gastrointestinal disorders) | 4 (13) | 5 (15) | 3 (9)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (45) | 8 (24) | 10 (28)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (17) | 6 (13) | 7 (17)
Death NOS (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (2) | 2 (4)
Fatigue (General disorders) | 1 (1) | 1 (1) | 3 (20)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (2) | 2 (2)
Weight gain (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 0 (0) | 4 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (12) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (16) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (6) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (10) | 3 (9) | 5 (12)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (5) | 2 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (14) | 2 (6) | 2 (3)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT03087708/Prot_SAP_000.pdf